CLINICAL TRIAL: NCT02224365
Title: Regular Apple Consumption Improves Cardiovascular Risk Factors and Glycemic Control in Overweight and Obese Prediabetics and Type 2 Diabetics
Brief Title: The Effects of Apple Consumption on Cardiovascular Health in Prediabetics and Type 2 Diabetics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: U.S. Apple Association (Unknown)
Responsible Party: Principal Investigator, Bahram Arjmandi, Margaret A. Sitton Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF02435; 2015.14930 (Other: FSU IRB)
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Cardiovascular Diseases; Prediabetes
Keywords: Diabetes; Arterial Stiffness; Blood Pressure; Endothelial Function; Body Composition; Glycemic Control; Apples; Functional Foods; Polyphenols; Fiber
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Prediabetic State

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apple (Experimental): 12 weeks of 75 g dried apple powder taken in 480 ml per day.
  Interventions: Dietary Supplement: Apple
- Placebo (Placebo Comparator): 12 weeks of 75 g apple-flavored placebo powder taken in 480 ml per day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Apple — 12 weeks of 75 g dried apple powder taken in 480 ml per day.
  Arms: Apple
Dietary Supplement: Placebo — 12 weeks of 75 g apple-flavored placebo powder taken in 480 ml per day.
  Arms: Placebo

SUMMARY:
The hypothesis of this study is that the daily consumption of 75 g dried apple powder for twelve weeks will improve arterial stiffness and blood pressure by improving endothelial-mediated vasodilation and vascular sympathetic activity and favorably altering biochemical markers associated with cardiovascular risk and glycemic control compared to a macronutrient-matched control powder. 50 men and women between the ages of 45 and 65 with prediabetes or type 2 diabetes who are overweight or obese will be included in the study. After a two-week run-in phase, eligible men and women will be randomly assigned to one of two treatment groups: 1) 75 g dried apple powder; or 2) 75 g placebo powder daily for twelve weeks. After an initial telephone screening, all participants will be requested to report to the study site for their first visit. On the first visit (screening), participants will be provided with verbal and written explanation of the project. They will then be asked to sign an informed consent form, followed by measuring fasting glucose levels and a medical history questionnaire to confirm prediabetes or type 2 diabetes. Baseline assessments will be performed for medical history, medication use, dietary intake, and physical activity. Qualified participants will be scheduled for their second visit two weeks later (actual baseline data collection) and randomly assigned to their treatment group. On the second (baseline) visit between the hours of 6:00-11:00 A.M., blood pressure and vascular function will be measured followed by blood draw and urine collection. Anthropometrics will be measured. Participants will be provided with their assigned treatment and will receive standard instructions on how to fill out daily diaries for their treatment, and for food and physical activity records. Blood pressure, vascular function, blood draw, urine collection, and anthropometric, body composition, diet, and physical activity assessments will be repeated at 6- (third visit), and 12-week (final visit) intervals. All cardiovascular measurements will be performed between 6:00 to 11:00 A.M., in a quiet temperature-controlled room in the supine position after an overnight fast and 12 hours after the abstinence of caffeine and/or 24 hours after the last bout of moderate to heavy physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (1 to 10 years postmenopausal)
* Aged 45-65 years
* Prediabetes or Type 2 Diabetes (Hemoglobin A1c ≥ 5.7%)
* Overweight or obese (body mass index between 25 and 40 kg/m2)

Exclusion Criteria:

* Diagnosed cardiovascular disease
* Uncontrolled hypertension (≥ 160/100 mmHg)
* Other active chronic diseases such as cancer, asthma, glaucoma, thyroid, kidney, liver and pancreatic disease
* Participating in a weight loss program
* Heavy smokers (> 20 cigarettes per day)
* Heavy drinkers (> 12 alcoholic drinks per week)
* Consumption of more than two apples per week
* Body mass index less than 25 or greater than 40 kg/m2)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 12 weeks
  By measuring brachial and aortic blood pressure at rest and during physiological stress (handgrip exercise and post-exercise muscle ischemia).

SECONDARY OUTCOMES:
Arterial Stiffness | 12 weeks
  By measuring arterial stiffness and augmentation index at rest and during physiological stress (handgrip exercise and post-exercise muscle ischemia).
Autonomic Control of Blood Pressure | 12 weeks
  By measuring blood pressure variability and baroreflex sensitivity at rest and during physiological stress.
Endothelial-mediated Vasodilation | 12 weeks
  By measuring flow-mediated dilation in the brachial artery.
Inflammation | 12 weeks
  By measuring markers of inflammation.
Oxidative Stress | 12 weeks
  By measuring markers of oxidative stress.
Insulin Sensitivity | 12 weeks
  By measuring fasting glucose, insulin, homeostatic model of insulin resistance, and hemoglobin A1C.
Atherogenic Markers | 12 weeks
  By measuring adhesion factors, lipid profiles, and atherogenic risk ratios.
Body Composition | 12 weeks
  By measuring fat mass and fat-free mass using dual-energy X-ray absorptiometry and anthropometrics.

CONTACTS AND LOCATIONS:
Overall Officials: Bahram H. Arjmandi, PhD, RD, Principal Investigator — Department of Nutrition, Food and Exercise Sciences, Center for Advancing Exercise and Nutrition Research on Aging, Florida State University; Arturo Figueroa, MD, PhD, Principal Investigator — Department of Nutrition, Food and Exercise Sciences, Florida State University; Sarah A. Johnson, PhD, RDN, Principal Investigator — Department of Food Science and Human Nutrition, Colorado State University
Locations (1):
- Department of Nutrition, Food and Exercise Sciences, Center for Advancing Exercise and Nutrition Research on Aging, Florida State University, Tallahassee, Florida, United States